CLINICAL TRIAL: NCT06813183
Title: Erzi̇ncan Binali Yildirim University
Brief Title: The Effect of Palmar Grip Reflex Stimulation on Pain During Heel Blood Collection in Newborns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Necla Kasımoğlu, Dr., Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123456
Record Dates: First submitted 2025-01-28; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pain
Keywords: palmar grasping reflex; newborn; nurse
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The heel prick attempt was planned one hour after the babies were breastfed (since the painful procedure may cause crying, doing it immediately after feeding may cause vomiting with crying).
  The infant included in the study in each group was placed in a resting period in his/her bed, undisturbed until 30 minutes before the start of the test (Dinç 2023). The heel prick procedure will be performed under radiant heater in the neonatal intensive care unit. The baby is monitored before starting the procedure under the radiant heater. Blood collection will be performed in accordance with the routine heel prick procedure.
  Physiologic parameters and pain levels 1 minute before (0 min), during, 2 and 5 min after the heel prick procedure in newborns in the NIPS control groups will be scored by the researcher and a second nurse with at least 5 years of experience in neonatal intensive care and recorded on the follow-up form (Çatal 2023).
  Interventions: Other: The palmar grasping reflex
- Experimental group (Experimental): In the experimental group, the baby is monitored under a radiant heater before the procedure. After the infant's initial physiologic parameters and NIPS are recorded, the palmar grasp reflex is stimulated just before the procedure begins. The palmar grasp reflex can be stimulated by moving an object distally across the palm of the hand. In newborns, the right hand is more dominant than the left hand in the palmar grasp reflex ( Fagard et al., 2017). The researcher will stimulate the palmar grasp reflex by moving the index finger distally along the palm of the infant's right hand. The reflex stimulation will be continued until the end of the 5th minute.
  Interventions: Other: The palmar grasping reflex

INTERVENTIONS:
Other: The palmar grasping reflex — In the experimental group, the baby is monitored under a radiant heater before the procedure. After the infant's initial physiologic parameters and NIPS are recorded, the palmar grasp reflex is stimulated just before the procedure begins. The palmar grasp reflex can be stimulated by moving an object distally across the palm of the hand. In newborns, the right hand is more dominant than the left hand in the palmar grasp reflex ( Fagard et al., 2017). The researcher will stimulate the palmar grasp reflex by moving the index finger distally along the palm of the infant's right hand. The reflex stimulation will be continued until the end of the 5th minute.
  Physiologic parameters will be scored by the investigator and a second nurse with at least 5 years of experience in neonatal intensive care and recorded on the follow-up form by scoring the pain levels 1 minute before (0 min), during, 2 and 5 min after the heel pricking procedure in the neonates in the NIPS intervention groups via the be
  Other Names: Experimental Procedure

SUMMARY:
Pain is defined by the International Association for the Study of Pain (IASP) as "an unpleasant sensory and emotional experience associated with or defined in terms of actual or potential tissue damage" . Since 1980, the newborn may encounter around 300 painful procedures with hospitalization. Before 1980, there was a misperception that newborns do not feel pain. Later research revealed that newborns feel pain and are sensitive to painful stimuli. Accurate assessment of pain in term or preterm newborns hospitalized in the Neonatal Intensive Care Unit (NICU) is of great importance in terms of mortality and morbidity due to the high prevalence of painful procedures, including daily procedural pain and postoperative pain.

An infant hospitalized in the neonatal intensive care unit for diagnosis and treatment purposes undergoes many interventions that cause pain and stress (intubation, arterial/venous catheter insertion, aspiration, chest tube, urinary catheter, nasogastric catheter insertion, dressing, plaster change, chest physiotherapy). Although newborns do not express pain verbally, they reveal pain with their reactions. Autonomic reactions in the body are understood from heart rate, respiration, and oxygen saturation. In addition to these, there are hormonal reactions. Behavioral responses include sleeping, waking up, crying, body movements and facial expressions.

Excessive, prolonged painful interventions in the newborn can have significant effects on adverse physiological, neuro-sensory, cognitive and behavioral health outcomes that can be life-threatening and have long-term effects on all major organ systems . It is stated that the neurodevelopment of infants exposed to repetitive painful interventional procedures may be negatively affected and may lead to problems such as sleep problems, attention deficit and learning disorders in later childhood. Therefore, it is important to reduce the stress caused by illness and hospitalization in newborns and minimize this traumatic effect.

Environmental (restricted noise and light) measures, sucrose solutions, kangaroo care, breast milk and breastfeeding, non-nutritive sucking, swaddling, massage, music, maternal (breast milk) and aromatic scents, positioning (developmental position), rocking and individualized developmental care have been shown to be effective in soothing infants during painful/stressful procedures.

The palmar grasping reflex is a component of attachment behavior that is considered therapeutic for both the infant and the caregiver. The grasping reflex is one of the most important primitive reflexes and is defined as an involuntary grasping and grasping movement in newborns. The grasping reflex occurs in both hands (palmar) and feet (plantar). The palmar grasp reflex is an involuntary flexion-adduction movement involving the hands and fingers. Holding and grasping the hand of the nurse, mother or caregiver can have a calming effect on the baby.

The Newborn Metabolic and Endocrine Disease Screening Program is implemented all over the world. The aim of the newborn screening program is to provide early diagnosis of congenital metabolic and endocrine disorders that may cause long-term sequelae or even result in death if left untreated. The metabolic diseases included in 13 newborn screening programs in Turkey are phenylketonuria (PKU), congenital hypothyroidism, biotinidase deficiency, cystic fibrosis (CF), congenital adrenal hyperplasia and spinal muscular atrophy (SMA).

Blood sample for newborn screening should ideally be taken at 36-72 hours. The application is performed by placing a few drops of blood taken from the heel of the baby's foot on Guthrie paper. Capillary blood is more easily collected and stored compared to whole blood or plasma samples. Therefore, capillary blood sample taken from the heel is preferred in the screening program. The medial (inner) or lateral (outer) parts of the plantar (sole) surfaces of the infant's heel should be used for blood collection. The heel of the baby's foot should be cleaned with 70% alcohol. Before piercing the skin, the alcohol should be allowed to dry so that the alcohol and blood do not mix. Mixing of blood and alcohol causes hemolysis of red blood cells and leads to erroneous results.

Although there are many studies on reducing and controlling the pain that newborns are exposed to in neonatal intensive care, the number of studies on the use of palmar grasping reflex during painful interventions is limited.

ELIGIBILITY:
The conditions sought for newborns included in the study are;

1. 38-42 weeks of gestation,
2. Within the first ten days of postnatal life,
3. 2500-4000 grams of birth weight,
4. Stable general condition,
5. Fed within an hour before the procedure,
6. Calm and not crying before the procedure,
7. 24-72 hours of postnatal age,
8. Newborns for whom one of the parents (mother or father) gave verbal and written consent will be included in the study.

Exclusion Criteria of the Study

* Newborns who need oxygen support,
* Are fed with an orogastric tube,
* Those whose first attempt at heel blood collection was unsuccessful,
* Those who need parenteral nutrition,
* Those receiving analgesic treatment,
* Those with physical, metabolic and genetic diseases,
* Those who have undergone a surgical procedure,
* Those with nerve damage or deformity in the extremity from which the heel blood will be collected,
* Newborns whose parents (mother or father) do not give verbal and written consent and wish to withdraw from the study will not be included.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | values 1 minute before, during, 2 and 5 minutes after the procedure during the interventions
  The Neonatal Infant Pain Scale (NIPS) is a scale that includes behavioral parameters used to assess the pain of premature and term newborns. The Neonatal Infant Pain Scale includes five behavioral parameters including facial expression, crying, arm and leg movements, and alertness, and a physiological parameter measurement in which respiration is evaluated. In the evaluation of the scale, the score varies between 0-7. In the scoring of the scale, 0-2 points indicate no pain/mild pain, 3-4 points indicate mild pain/moderate pain and >4 points indicate severe pain. Cronbach's alpha coefficient of the scale was 0.95 before the procedure, 0.87 during the procedure and 0.88 after the procedure (Lawrence, 1993). Turkish validity and reliability of the scale was performed by Akdovan et al. (1999).

SECONDARY OUTCOMES:
Newborn' s SpO2 | values 1 minute before, during, 2 and 5 minutes after the procedure during the interventions
  This form was developed by the researchers in line with the literature in order to record information such as physiologic parameters of newborns (SpO2, heart rate), crying time and procedure time (Çatal 2023).
Newborn' s hearth rate | values 1 minute before, during, 2 and 5 minutes after the procedure during the interventions
  This form was developed by the researchers in line with the literature in order to record
Newborn' s crying time | values 1 minute before, during, 2 and 5 minutes after the procedure during the interventions
  This form was developed by the researchers in line with the literature in order to record

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yıldırım University, Merkez, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No